CLINICAL TRIAL: NCT06374641
Title: The Effects of a Novel Mitochondrial Substrate Supplement on Exercise Performance and Cognitive Function
Acronym: MCh1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Mitocholine Ltd (Industry); Innovate UK (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 5514255
Record Dates: First submitted 2024-03-12; First posted 2024-04-18 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Exercise Performance; Cognitive Function
Keywords: choline; nicotinamide; succinate; supplement; exercise; cognitive function
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Trials will be randomised and counterbalanced to remove any trial-order effect.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Partners Innovate UK and Mitocholine Ltd will also be masked. Masking will be performed by an individual outside of the research group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mitochondrial Substrate Supplement then Placebo (Experimental): Administered as a drink, participants receive mitochondrial substrate supplement to be taken in the morning in a fasted state in a dose of 65 mL/day twice daily for 16 days. After a washout period of 28 (or 46 for young females) days they then receive the placebo matching the mitochondrial substrate supplement to be taken in the same way, for 16 days.
  Each 65 mL dose of the supplement provides a dose of 481.66 mg choline, 273.01 mg succinic acid, and 15 mg nicotinamide. 65 mL of placebo consists of Aspartame (15.3 mg), Acesulfame-K (10.3 mg), Potassium Sorbate (9.1 mg), Sodium Benzoate (9.8 mg), Cellulose Gum (6.5 mg), Gluconic acid (1105.0 mg), Ginger Natural Flavouring (130.0 mg), Orange Natural Flavouring (130.0 mg), Bitter Sensation Natural Flavouring (65.0 mg), Natural Colour (colouring food) (26.0 mg), Water (63493.0 mg).
  Interventions: Dietary Supplement: Mitochondrial Substrate Supplement; Dietary Supplement: Placebo Supplement
- Placebo then Mitochondrial Substrate Supplement (Placebo Comparator): Administered as a drink, participants receive placebo supplement matching the mitochondrial substrate supplement in taste and appearance, to be taken in a dose of 65 mL twice daily for 16 days. After a washout period of 28 (or 46 for young females) days they then receive the mitochondrial substrate supplement, to be taken in the same way, for 16 days.
  Each 65 mL dose of the placebo supplement provides 481.66 mg choline, 273.01 mg succinic acid, and 15 mg nicotinamide. 65 mL of placebo consists of Aspartame (15.3 mg), Acesulfame-K (10.3 mg), Potassium Sorbate (9.1 mg), Sodium Benzoate (9.8 mg), Cellulose Gum (6.5 mg), Gluconic acid (1105.0 mg), Ginger Natural Flavouring (130.0 mg), Orange Natural Flavouring (130.0 mg), Bitter Sensation Natural Flavouring (65.0 mg), Natural Colour (colouring food) (26.0 mg), Water (63493.0 mg).
  Interventions: Dietary Supplement: Mitochondrial Substrate Supplement; Dietary Supplement: Placebo Supplement

INTERVENTIONS:
Dietary Supplement: Mitochondrial Substrate Supplement — Mitochondrial Substrate supplement, 2xdaily 65 mL drink
  Other Names: Mitocholine, MiBrain
Dietary Supplement: Placebo Supplement — Placebo supplement, 2xdaily 65 mL drink

SUMMARY:
The goal of this clinical trial is to compare the effects of taking a new supplement for 16 days on cognitive function and exercise performance, compared to a placebo (a supplement that looks and tastes the same, but doesn't have the same ingredients) in 40 healthy individuals - 20 young individuals (aged 18-30) and 20 older individuals (aged 50-65).

The main questions it aims to answer are:

* If taking the supplement for 16 days improves exercise performance, or the speed with which the body responds to the commencement of exercise.
* If taking the supplement improves cognitive function.

Participants will visit the lab on 5 separate occasions to:

* complete some cognitive tests
* complete exercise performance tests
* provide blood samples

All exercise tests will be on an exercise bike.

After 28 (or 46 for pre-menopausal females) days to make sure the supplement has left the body fully, participants will consume the opposite supplement and repeat the tests.

DETAILED DESCRIPTION:
This study is a randomised, placebo-controlled, cross-over trial investigating the effects of supplementing with a novel mitochondrial substrate supplement on exercise performance and cognitive function.

The supplement is composed of three bioactive components: choline, nicotinamide and succinate. All three components are available on the market as supplements and/or as food additives, but have not previously been combined.

This study will recruit 40 individuals in two cohorts. The first cohort will consist of 20 young individuals (aged 18-30) and the second cohort will consist of 20 older individuals (aged 50-65). Individuals will be block randomised into two groups within each cohort, taking either the placebo or supplement first. Trials will be counterbalanced by Latin square to remove any trial-order effect.

This study will involve 5 lab visits per participant, including a familiarisation visit and a further 2 visits per trial arm. Familiarisation will consist of questionnaires and cognitive tests, warm-up and ramp incremental test on a cycle ergometer for all participants. The ramp incremental test will commence with a 3-minute unloaded baseline period followed by an increase in work rate until task failure. Task failure will be defined as a drop by >10 rpm below participants' self-selected cadence (which is expected to lie between 70 and 100 rpm). Following a rest period, participants in the 'young' cohort will also complete a 3-minute all-out test on a cycle ergometer.

Participants will be supplemented with 65 mL.d-1 of either a placebo or the supplement twice daily for 16 days while recording food intake and exercise activities. On days 15 and 16 of supplementation, participants will return to the lab for testing. Testing on day 15 will consist of questionnaires and cognitive tests, a venous blood sample, and a 3-minute all out test (young cohort) or ramp incremental test (older cohort) on a cycle ergometer. Venous samples will be collected prior to exercise.

Testing on day 16 will consist of a series of three 6-min step tests, from unloaded to moderate intensity, with a 15-minute rest period between each test. Moderate exercise is defined as exercise which occurs below the lactate threshold. Participants will then complete an intermittent exercise protocol consisting of alternating 60-second periods of severe intensity exercise and 30-second periods of recovery until they reach the limit of tolerance. Severe intensity is defined as exercise which occurs above the critical power, where VO2max is reached at exhaustion. All tests will be conducted on a cycle ergometer.

Following completion of the first trial arm, participants will undergo a 28 or 46 (pre-menopausal females) day washout period. The washout period for young female participants is adjusted to enable all testing to occur in the same phase of the menstrual cycle and thus remove potential associated confounding effects. Participants will then repeat the supplementation protocol and testing visits on days 15 and 16 with the opposing supplement.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be deemed eligible to participate provided they are willing and able to follow the study instructions and

  1. are able to take part in intense exercise (as assessed via Physical Activity Readiness Questionnaire (PARQ))
  2. are able to consume a dietary supplement
  3. are not overweight/obese (assessed by BMI)
  4. do not have any cardiovascular, respiratory, metabolic or musculoskeletal disorders, or any other contraindication to the performance of maximal exercise.

Exclusion Criteria:

1. Aged 31-49 and aged 66+.
2. underlying illness or injury (assessed via PARQ)
3. overweight or obese individuals (BMI of >30 kg.m-2).
4. Cardiovascular, respiratory, metabolic or musculoskeletal disorders (assessed by screening form).
5. Use of dietary supplements, tobacco smoking.
6. Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Exercise Capacity | Day 15 and 16
  Exercise performance as measured by ramp incremental test (older group) or 3 minute all out test (young group) and intermittent exercise test. The ramp incremental cycling test is well-established for the determination of maximal oxygen uptake (VO2max) and gaseous exchange threshold, which are key markers of cardiorespiratory health and predictor of endurance exercise performance. The 3 minute all out test is commonly used to determine critical power and W'. The critical power represents the highest power output an individual can sustain while remaining in an aerobic steady state, and the W' represents the anaerobic capacity.
  The intermittent test consists of intermittent exercise in which 1 min of severe intensity exercise is alternated with 30 s of lower intensity exercise until the participant reaches their limit of tolerance. Time to exhaustion allows for assessment of exercise capacity.
VO2 kinetic response to exercise | Day 16
  The VO2 response measured during step test from unloaded to moderate intensity exercise. The participant will cycle against a low resistance and then the resistance on the pedals will be increased abruptly to provide a moderate-intensity work rate which will be maintained for 6 minutes. The VO2 response will then be examined from the onset of exercise to the attainment of a steady state. The VO2 responses to the three step tests will be averaged and modelled to provide information on the rate at which the muscle mitochondria use oxygen to supply energy to meet the demands of the exercise. The steady-state VO2 value for the imposed work rate also allows for the assessment of exercise economy.
Cognitive Function (Stroop test) | Day 15
  Cognitive function tested via Stroop test administered by computerised system.
Cognitive Function (decision reaction test) | Day 15
  Cognitive function tested via decision reaction test administered by computerised system.
Grip Strength | Day 15
  Grip strength measured by hand strength dynamometer.

SECONDARY OUTCOMES:
Capillary Blood Lactate | Before and after each step during the step test, and before and after every 2 exercise bouts during the intermittent exercise protocol.
  Capillary Blood Lactate used during step tests and intermittent exercise tests to examine the production of lactate and inferred levels of muscle acidosis.
Questionnaire 1 | Day 16
  To assess participant experience during the supplementation period and study protocol with regard to factors such as fatigue, stress, sleep and perceived effort.
Questionnaire 2 | Day 15
  To assess participant experience of the supplement with regard to factors such as perceived effects, tolerance and taste.
Venous Blood [Betaine] | Day 15
  Assessment of Venous Blood [Betaine].
Venous Blood [Choline] | Day 15
  Assessment of Venous Blood [Choline].
Venous blood [S-Adenosyl methionine] | Day 15
  Assessment of Venous Blood [S-Adenosyl methionine].
Venous blood [glucose]. | Day 15
  Assessment of Venous Blood [glucose].
Venous blood [insulin]. | Day 15
  Assessment of Venous Blood [insulin].
Venous blood [trimethylamine N-oxide]. | Day 15
  Assessment of Venous Blood [triglycerides].

CONTACTS AND LOCATIONS:
Overall Officials: Andy M Jones, PhD, DSc, Principal Investigator — University of Exeter
Locations (1):
- Richards Building St. Lukes Campus University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available as anonymised data sets of final published data in supplementary material of publications associated with this study.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available on completion of data collection and analysis. Data will be available without an end date.
Access Criteria: Data will be available in supplementary material for publications resulting from this study, and following requests from fellow researchers.

REFERENCES:
- [Result] Vanhatalo A, Doust JH, Burnley M. Determination of critical power using a 3-min all-out cycling test. Med Sci Sports Exerc. 2007 Mar;39(3):548-55. doi: 10.1249/mss.0b013e31802dd3e6. PMID 17473782
- [Result] Bailey SJ, Winyard P, Vanhatalo A, Blackwell JR, Dimenna FJ, Wilkerson DP, Tarr J, Benjamin N, Jones AM. Dietary nitrate supplementation reduces the O2 cost of low-intensity exercise and enhances tolerance to high-intensity exercise in humans. J Appl Physiol (1985). 2009 Oct;107(4):1144-55. doi: 10.1152/japplphysiol.00722.2009. Epub 2009 Aug 6. PMID 19661447
- [Result] Chidnok W, Dimenna FJ, Bailey SJ, Vanhatalo A, Morton RH, Wilkerson DP, Jones AM. Exercise tolerance in intermittent cycling: application of the critical power concept. Med Sci Sports Exerc. 2012 May;44(5):966-76. doi: 10.1249/MSS.0b013e31823ea28a. PMID 22033512